CLINICAL TRIAL: NCT00056472
Title: Effectiveness of Selective Serotonin Reuptake Inhibitors Combined With Antipsychotic Medication for the Treatment of Psychotic Depression
Brief Title: Study of Pharmacotherapy of Psychotic Depression
Acronym: STOP-PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01MH062624 (NIH); U01MH062624 (NIH); U01MH062565 (NIH); U01MH062518 (NIH); U01MH062446 (NIH)
Record Dates: First submitted 2003-03-14; First posted 2003-03-17 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-06

CONDITIONS: Major Depressive Disorder With Psychotic Features
Keywords: Major depressive disorder with psychotic features; Delusional Depression; Randomized Trial; Combination Treatment; SSRI; Atypical Antipsychotic
MeSH Terms: interventions — Olanzapine; Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- olanzapine/sertraline combination (Active Comparator): sertraline plus olanzapine
  Interventions: Drug: Olanzapine; Drug: Sertraline
- olanzapine plus placebo (Placebo Comparator): olanzapine (5 - 20mg/day) plus placebo
  Interventions: Drug: Olanzapine; Other: placebo

INTERVENTIONS:
Drug: Olanzapine — 10-20mg/day
  Other Names: Zyprexa
Drug: Sertraline — 150-200mg/day
  Other Names: Zoloft
  Arms: olanzapine/sertraline combination
Other: placebo — tablet that ressembles sertraline but contains no medication
  Arms: olanzapine plus placebo

SUMMARY:
This study will determine the effectiveness of combining selective serotonin reuptake inhibitors (SSRIs) with antipsychotic medications in the treatment of psychotic depression.

DETAILED DESCRIPTION:
Approximately 25% of people who are admitted to hospitals for depression suffer from psychotic depression. People with psychotic depression experience hallucinations,and, more commonly delusions, in addition to major depression. Psychotic experiences may be either congruent with the theme of depression or incongruent, without an apparent relationship to feeling depressed. This study will determine the effectiveness of combining a selective serotonin reuptake inhibitor (SSRI) with antipsychotic medication in the treatment of psychotic depression accompanied by at least one identifiable delusion. The study will also evaluate the difference in treatment response of young adults versus geriatric patients.

This double-blind study will last a total of 12 weeks. Participants will be randomly assigned to receive either olanzapine, an atypical antipsychotic drug, combined with sertraline, an SSRI, or olanzapine alone. Following baseline assessments, study visits will occur weekly until Week 6, and then bi-weekly until Week 12. Participants who do not respond to either treatment may leave the study at any time. Participants who achieve either partial or full response may participate in an additional 20-week study.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder, single or recurrent, with psychotic features

Exclusion Criteria:

* History of substance abuse or dependence within the 3 months prior to enrollment
* Acute or unstable medical illness
* Diagnosis of schizophrenia or other psychotic disorders
* Pregnant
* Intolerance to SSRIs or olanzapine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2003-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barnett Meyers, MD, Principal Investigator — Cornell University
Locations (4):
- United States (3):
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Cornell University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kruizinga J, Liemburg E, Burger H, Cipriani A, Geddes J, Robertson L, Vogelaar B, Nolen WA. Pharmacological treatment for psychotic depression. Cochrane Database Syst Rev. 2021 Dec 7;12(12):CD004044. doi: 10.1002/14651858.CD004044.pub5. PMID 34875106
- [Derived] Bingham KS, Meyers BS, Mulsant BH, Rothschild AJ, Whyte EM, Banerjee S, Artis AS, Alexopoulos GS, Flint AJ; STOP-PD Study Group. Stabilization treatment of remitted psychotic depression: the STOP-PD study. Acta Psychiatr Scand. 2018 Sep;138(3):267-273. doi: 10.1111/acps.12937. Epub 2018 Jun 29. PMID 29959765
- [Derived] Bingham KS, Rothschild AJ, Mulsant BH, Whyte EM, Meyers BS, Banerjee S, Szanto K, Flint AJ; STOP-PD Study Group. The Association of Baseline Suicidality With Treatment Outcome in Psychotic Depression. J Clin Psychiatry. 2017 Sep/Oct;78(8):1149-1154. doi: 10.4088/JCP.16m10881. PMID 28445632
- [Derived] Gerretsen P, Flint AJ, Whyte EM, Rothschild AJ, Meyers BS, Mulsant BH. Impaired insight into delusions predicts treatment outcome during a randomized controlled trial for Psychotic Depression (STOP-PD study). J Clin Psychiatry. 2015 Apr;76(4):427-33. doi: 10.4088/JCP.14m09003. PMID 25919834
- [Derived] Deligiannidis KM, Rothschild AJ, Barton BA, Kroll-Desrosiers AR, Meyers BS, Flint AJ, Whyte EM, Mulsant BH; STOP-PD Study Group. A gender analysis of the study of pharmacotherapy of psychotic depression (STOP-PD): gender and age as predictors of response and treatment-associated changes in body mass index and metabolic measures. J Clin Psychiatry. 2013 Oct;74(10):1003-9. doi: 10.4088/JCP.13m08400. PMID 24229753
- [Derived] Ostergaard SD, Meyers BS, Flint AJ, Mulsant BH, Whyte EM, Ulbricht CM, Bech P, Rothschild AJ; STOP-PD Study Group. Measuring psychotic depression. Acta Psychiatr Scand. 2014 Mar;129(3):211-20. doi: 10.1111/acps.12165. Epub 2013 Jun 25. PMID 23799875
- [Derived] Flint AJ, Iaboni A, Mulsant BH, Rothschild AJ, Whyte EM, Meyers BS; STOP-PD Study Group. Effect of sertraline on risk of falling in older adults with psychotic depression on olanzapine: results of a randomized placebo-controlled trial. Am J Geriatr Psychiatry. 2014 Apr;22(4):332-6. doi: 10.1016/j.jagp.2013.01.067. Epub 2013 May 2. PMID 23642462
- [Derived] Blumberger DM, Mulsant BH, Kanellopoulos D, Whyte EM, Rothschild AJ, Flint AJ, Meyers BS. The incidence of tardive dyskinesia in the study of pharmacotherapy for psychotic depression. J Clin Psychopharmacol. 2013 Jun;33(3):391-7. doi: 10.1097/JCP.0b013e31828bf059. PMID 23609383
- [Derived] Weissman J, Flint A, Meyers B, Ghosh S, Mulsant B, Rothschild A, Whyte E; STOP-PD Study Group. Factors associated with non-completion in a double-blind randomized controlled trial of olanzapine plus sertraline versus olanzapine plus placebo for psychotic depression. Psychiatry Res. 2012 May 30;197(3):221-6. doi: 10.1016/j.psychres.2012.02.015. Epub 2012 Mar 31. PMID 22464991
- [Derived] Meyers BS, Flint AJ, Rothschild AJ, Mulsant BH, Whyte EM, Peasley-Miklus C, Papademetriou E, Leon AC, Heo M; STOP-PD Group. A double-blind randomized controlled trial of olanzapine plus sertraline vs olanzapine plus placebo for psychotic depression: the study of pharmacotherapy of psychotic depression (STOP-PD). Arch Gen Psychiatry. 2009 Aug;66(8):838-47. doi: 10.1001/archgenpsychiatry.2009.79. PMID 19652123
- [Derived] Schaffer A, Flint AJ, Smith E, Rothschild AJ, Mulsant BH, Szanto K, Peasley-Miklus C, Heo M, Papademetriou E, Meyers BS. Correlates of suicidality among patients with psychotic depression. Suicide Life Threat Behav. 2008 Aug;38(4):403-14. doi: 10.1521/suli.2008.38.4.403. PMID 18724788
- [Derived] Smith E, Rothschild AJ, Heo M, Peasley-Miklus C, Caswell M, Papademetriou E, Flint AJ, Mulsant BH, Meyers BS; STOP-PD Collaborative Study Group. Weight gain during olanzapine treatment for psychotic depression: effects of dose and age. Int Clin Psychopharmacol. 2008 May;23(3):130-7. doi: 10.1097/YIC.0b013e3282f424d6. PMID 18408527
- [Derived] Rothschild AJ, Winer J, Flint AJ, Mulsant BH, Whyte EM, Heo M, Fratoni S, Gabriele M, Kasapinovic S, Meyers BS; Study of Pharmacotherapy of Psychotic Depression (STOP-PD) Collaborative Study Group. Missed diagnosis of psychotic depression at 4 academic medical centers. J Clin Psychiatry. 2008 Aug;69(8):1293-6. doi: 10.4088/jcp.v69n0813. PMID 18384244
- [Derived] Andreescu C, Mulsant BH, Peasley-Miklus C, Rothschild AJ, Flint AJ, Heo M, Caswell M, Whyte EM, Meyers BS; STOP-PD Study Group. Persisting low use of antipsychotics in the treatment of major depressive disorder with psychotic features. J Clin Psychiatry. 2007 Feb;68(2):194-200. doi: 10.4088/jcp.v68n0203. PMID 17335316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the inpatient and outpatient services of four academic sites between December of 2002 and June of 2007.
Pre-assignment Details: Antidepressant and antipsychotic medications being taken at entry were tapered and discontinued prior to randomization. Consented subjects were required to meet criteria for unipolar major depression and have at least one delusion. Subjects were also excluded if an unstable medical condition or evidence of recent substance abuse were present.
Groups:
- Sertraline Plus Olanzapine: 50-200mg/day sertraline plus 5-20mg/day olanzapine
- Olanzapine Plus Placebo: 5-20mg/day olanzapine plus placebo
Period: Overall Study
Arm/Group | Sertraline Plus Olanzapine | Olanzapine Plus Placebo
Started | 129 | 130
Completed | 81 | 61
Not Completed | 48 | 69

BASELINE CHARACTERISTICS:
Groups:
- Pharmacotherapy: sertraline plus olanzapine
- Monotherapy: placebo plus olanzapine
- Total: Total of all reporting groups
Arm/Group | Pharmacotherapy | Monotherapy | Total
Number analyzed (Participants) | 129 | 130 | 259
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 77 | 73 | 150
  >=65 years | 52 | 56 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 83 | 166
  Male | 46 | 47 | 93
Region of Enrollment [Number; unit: participants]
  United States | 89 | 89 | 178
  Canada | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Remission of Depression Hamilton Depression Scale (Ham-D) and Psychosis Schedule for Affective Disorders in Schizophrenia - Delusional Item (SADS) During the Course of the Trial
Description: Remission was defined as scores on Ham-D of less than 10 at two consecutive assessments and the absence of delusions (measured as SADS delusional item scores of 1) at the second assessment of the two-assessment remission of depression interval.
  Scores on Ham-D range from 0 to 52 with higher scores indicating more severe depression. Scores on SADS range from 1 to 7 with higher scores indicating the delusions(s) more adversely effect the subject's behavior.
Time Frame: Weeks 1 to 12
Measure: Number; unit: participants
Arm/Group | Pharmacotherapy | Monotherapy
Number analyzed (Participants) | 124 | 126
participants | 54 | 31
Statistical Analysis 1: Comparison: Pharmacotherapy vs Monotherapy; Predicting remission rates of 40% in combination therapy and 20% in monotherapy subjects, 260 subjects randomized into the two treatment groups would provide >80% power at a two-tailed alpha level of .05. Treatment efficacy was compared between groups based on intent-to-treat analyses for the longitudinal binary outcome of remission using mixed effects logistic regression with a random intercept that included treatment and time as fixed effects and a treatment by time interaction effect; Test type: Superiority or Other; p < .001, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI [1.12 to 1.47]

2. Secondary Outcome: Scores on CGI-S Compared to Baseline Over the Course of the Trial
Description: A measure of overall symptom severity, the Clinical Global Impressions, Severity of Illness Scale (CGI-S). It is a seven point scale with a one indicating not at all ill, and seven indicating the most extremely ill. This rating was done each week after baseline by the PI at each site after visiting with the patient.
Time Frame: Weeks 1 to 12
Measure: Mean (Standard Error); unit: units on CGI scale
Arm/Group | Pharmacotherapy | Monotherapy
Number analyzed (Participants) | 124 | 126
units on CGI scale | 2.24 (.07) | 2.48 (.07)
Statistical Analysis 1: Comparison: Pharmacotherapy vs Monotherapy; Intent-to-treat changes in global improvement from week to week compared to baseline (CGI-S) over the course of the trial using longitudinal mixed effects linear regression models. The null hypothesis is that there is no difference in overall change in CGI-S; Test type: Superiority or Other; p = .02, Mixed Models Analysis — The p-value is for the overall mean CGI-S score compared to baseline; This was a longitudinal analysis of CGI-S scores compared to baseline

3. Other Pre Specified Outcome: Mean Score Hamilton Depression Rating Scale (Ham-D) Over the Course of the Trial From Week to Week.
Description: The Ham-D measures depression severity. Scores on Ham-D range from 0 to 52 with higher scores indicating more severe depression.
Time Frame: Weeks 1 to 12
Measure: Mean (Standard Error); unit: Scores on Ham-D
Arm/Group | Pharmacotherapy | Monotherapy
Number analyzed (Participants) | 124 | 125
Scores on Ham-D | 13.27 (.61) | 16.63 (.61)
Statistical Analysis 1: Comparison: Pharmacotherapy vs Monotherapy; Intent-to-treat between group comparison using longitudinal mixed effects regression; Test type: Superiority or Other; p < .001, Mixed Models Analysis — The p-value is for the overall mean across all time points between each treatment group

ADVERSE EVENTS:
Time Frame: Subjects participated for a maximum of 12 weeks. Study duration of 4.5 years
Description: Extrapyramidal symptoms assessed using the Simpson Angus Scale, incident akathisia using the Barnes Akathisia Scale and tardive dyskinesia was assessed using the Abnormal Involuntary Movement Scale. Changes in UKU measured at each visit. Metabolic labs assessed monthly. Attrition. Other adverse events self-reported throughout study participation.
Arm/Group | Pharmacotherapy | Monotherapy
Serious Adverse Events (participants affected / at risk) | 9/129 | 3/130
Other Adverse Events (participants affected / at risk) | 39/129 | 35/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pharmacotherapy (N=129) | Monotherapy (N=130)
worsening depression (Psychiatric disorders) | 9 | 3 — worsening symptoms of depression requiring (re)hospitalization
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
broken hip (Musculoskeletal and connective tissue disorders) | 1 | 0
knee sepsis (Musculoskeletal and connective tissue disorders) | 0 | 1
chest pain (Vascular disorders) | 0 | 1
accidental overdose (General disorders) | 0 | 1
leg pain/edema (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pharmacotherapy (N=129) | Monotherapy (N=130)
weight gain (Metabolism and nutrition disorders) | 39 | 35
fall (General disorders) | 25 | 16
sleepiness/sedation (General disorders) | 9 | 11
increased lab values (Metabolism and nutrition disorders) | 14 | 3 — triglycerides, cholesterol, LFTs
reduced sleep (General disorders) | 4 | 7
pedal edema/edema (Vascular disorders) | 7 | 2
Increased fatigability (General disorders) | 2 | 7
increased sleep (General disorders) | 4 | 4
increased dream activity (General disorders) | 7 | 1
constipation (Gastrointestinal disorders) | 3 | 4
dizziness/feeling faint (General disorders) | 5 | 2
akathisia (Nervous system disorders) | 0 | 7
nausea/vomiting (Gastrointestinal disorders) | 2 | 4
tremor (Nervous system disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No